CLINICAL TRIAL: NCT06215534
Title: Determination of the Postprandial Glycemic Response and Glycemic Index of Nutritional Products: A Randomized Controlled Clinical Trial in Healthy Individuals
Brief Title: Glin3: Assessment of the Glycemic Responses to Nutritional Products
Acronym: GLIN#3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23REX0060928
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Glycemic Response
Keywords: Glycemic response; Glycemic Index; Nutritional products; Healthy individuals

STUDY DESIGN:
Intervention Model Description: 12 products will be tested (2 x 6 products + each 3 contls) that means 18 ärms"in total
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- arm 1 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: first reference product series 1
- arm 2 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: second reference product seies 1
- arm 3 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: third reference product series 1
- arm 4 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: first concept product series 1
- arm 5 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: second concept product series 1
- arm 6 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: third concept product series 1
- arm 7 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 4th concept product seris 1
- arm 8 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 5th concept product series 1
- arm 9 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 6th concept product series 1
- arm 10 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 1st reference product series 2
- arm 11 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 2nd reference product series 2
- arm 12 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 3rd reference product series 2
- arm 13 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 1st concept product series 2
- arm 14 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 2nd concept product series 2
- arm 15 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 3rd concept product series 2
- arm 16 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 4th concept product series 2
- arm 17 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 5th concept product series 2
- arm 18 (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: 6th concept product series 2

INTERVENTIONS:
Dietary Supplement: first reference product series 1 — dextrose (containing 25 grams of carbohydrates)
  Arms: arm 1
Dietary Supplement: second reference product seies 1 — dextrose (containing 25 grams of carbohydrates)
  Arms: arm 2
Dietary Supplement: third reference product series 1 — dextrose (containing 25 grams of carbohydrates)
  Arms: arm 3
Dietary Supplement: first concept product series 1 — Standard tube feed (containing 25 grams of carbohydrates)
  Arms: arm 4
Dietary Supplement: second concept product series 1 — Tube feed with added fibers (containing 25 grams of carbohydrates)
  Arms: arm 5
Dietary Supplement: third concept product series 1 — Tube feed with extra energy (containing 25 grams of carbohydrates)
  Arms: arm 6
Dietary Supplement: 4th concept product seris 1 — Tube feed with extra energy and added fibers (containing 25 grams of carbohydrates)
  Arms: arm 7
Dietary Supplement: 5th concept product series 1 — Plant based oral nutritional supplement for disease related malnutrition (containing 25 grams of carbohydrates
  Arms: arm 8
Dietary Supplement: 6th concept product series 1 — Oral nutritional supplement for disease related malnutrition in patients with malabsorption and/or maldigestion (containing 25 grams of carbohydrates
  Arms: arm 9
Dietary Supplement: 1st reference product series 2 — dextrose (containing 25 grams of carbohydrates)
  Arms: arm 10
Dietary Supplement: 2nd reference product series 2 — dextrose (containing 25 grams of carbohydrates)
  Arms: arm 11
Dietary Supplement: 3rd reference product series 2 — dextrose (containing 25 grams of carbohydrates)
  Arms: arm 12
Dietary Supplement: 1st concept product series 2 — High energy plant based tube feed (containing 25 grams of carbohydrates)
  Arms: arm 13
Dietary Supplement: 2nd concept product series 2 — High energy plant based tube feed with added fibers (containing 25 grams of carbohydrates)
  Arms: arm 14
Dietary Supplement: 3rd concept product series 2 — High protein tube feed (containing 25 grams of carbohydrates)
  Arms: arm 15
Dietary Supplement: 4th concept product series 2 — High protein, high energy tube feed based on peptides (containing 25 grams of carbohydrates)
  Arms: arm 16
Dietary Supplement: 5th concept product series 2 — Oral nutritional supplement for disease related malnutrition in patients with muscle loss (containing 25 grams of carbohydrates)
  Arms: arm 17
Dietary Supplement: 6th concept product series 2 — Oral nutritional supplement for disease related malnutrition (containing 25 grams of carbohydrates)
  Arms: arm 18

SUMMARY:
This study assesses the glycemic responses to nutritional products. During a study visit fasted subjects will consume one serving of the reference product or the test product. Capillary blood samples will be taken at baseline and at several time-points over a 2-hr period. Several nutritional products will be tested over time.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 65 years
* Body mass index (BMI) between 18.5 and 27 kg/m²

Exclusion Criteria:

* Baseline fasting Glucose ≥6.1 at screening visit
* Known history of gastrointestinal disease, bariatric surgery, AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), or any condition which might, in the opinion of the medical director either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Use of medications known to influence carbohydrate metabolism, gastrointestinal function or appetite, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or any medication which might, in the opinion of the medical director either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or surgical event within 3 months of screening.
* Known intolerance, sensitivity or allergy to test products.
* Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
* History of cancer in the prior two years, except for non-melanoma skin cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
The glycemic index of nutritional products | 6 months

SECONDARY OUTCOMES:
1. The postprandial glucose levels at each time point after each test product compared with the mean of the 3 references | 6 months
2. The postprandial incremental area under the curve (iAUC) after each test product compared with the mean of the 3 references | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Inquis Clinical research, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No